CLINICAL TRIAL: NCT05893004
Title: German Translation and Cross-cultural Adaptation of the Headache Screening Questionnaire (HSQ) Followed by a Test-retest Reliability Study.
Acronym: GUR-HSQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Markus J. Ernst (Other)
Responsible Party: Sponsor-Investigator, Markus J. Ernst, Phd., Zurich University of Applied Sciences
Organization: Zurich University of Applied Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GUR-HSQ
Record Dates: First submitted 2023-05-28; First posted 2023-06-07 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Migraine; Tension-Type Headache
MeSH Terms: conditions — Migraine Disorders; Tension-Type Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test-Retest (Experimental): sample of convenience headache suffereres will be tested twice
  Interventions: Diagnostic Test: Headache Screening Questionnaire

INTERVENTIONS:
Diagnostic Test: Headache Screening Questionnaire — The Dutch Headache Screening Questionnaire (HSQ) is the only screening questionnaire based on ICHD-3 which has at least moderate confidence in its criterion validity according to GRADE. The HSQ has already been translated into Portuguese and validated5. The HSQ has only 8 items and requires little time to complete. Due to its good sensitivity, the HSQ screening questionnaire is particularly well suited to exclude migraine.

SUMMARY:
The goal of this study is to learn more about the Headache Screening Questionnaire in people with Headache. The main question is:

Does the lower limit of a 95% confidence interval of the HSQ in physiotherapy during a period of 2 to 4 weeks reach at least 0.4?

DETAILED DESCRIPTION:
Data are collected using the REDCap web application (https://redcap.zhaw.ch/). REDCap is designed for the creation and administration of online surveys. Respondents can access the survey directly via a QR code or link and complete the screening questionnaire via smartphone or computer. In a first step, the participating persons are included or excluded based on the criteria mentioned (chapter: Proband:innen). Once eligibility has been confirmed, the HSQ is completed online for the first time in a second step. After that, the test persons will receive a reminder e-mail after 2 weeks to complete the retest online. After the reminder email the test persons have 2 weeks to complete the retest. Those who participate later will be excluded and not included in the data analysis. In addition, the retest asks whether the headaches have changed compared to the test due to the physiotherapeutic treatment. This is asked with a three Likert scale (not changed, slightly changed, strongly changed). The severely changed headaches are not included in the analysis.

Translated with www.DeepL.com/Translator (free version)

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are older than 18 years,
* live in Switzerland
* speak and understand German
* have had multiple headache episodes of the same or similar type

Exclusion Criteria:

* individuals with other known neurological conditions,
* known cognitive impairment
* known secondary headache types

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Kappe Value | Participants are assessed based on criteria (chapter: participants). Eligible individuals complete the HSQ online. A reminder email is sent after 2 weeks for the retest. Participants have 2 weeks to complete it. Late participants are excluded from analys
  The HSQ uses nominal variables for screening the two primary headaches with defined cut-offs of 6 and 8 points for migraine and TTH, respectively. Therefore, for the test-retest reliability analysis, a Cohen's kappa with corresponding 95% confidence interval is calculated for both migraine and TTH.

CONTACTS AND LOCATIONS:
Overall Officials: Markus J Ernst, MSc, Study Director — Zurich University of Applied Sciences
Locations (1):
- Zurich University of applied sciences, Winterthur, Switzerland